CLINICAL TRIAL: NCT04472832
Title: A Phase 1, Randomized, Four-Period, Crossover Food-Effect Study With Mitapivat Sulfate In Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Mitapivat (AG-348) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AG348-C-014
Record Dates: First submitted 2020-07-13; First posted 2020-07-15 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — mitapivat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Placebo Comparator): Participants will receive a single oral dose of mitapivat-matching placebo under fasted conditions on Day 1 of each of 4 periods.
  Interventions: Drug: Placebo for Treatment A
- Treatment B (Experimental): Participants will receive a single oral dose of mitapivat 100 milligrams (mg) and placebo under fasted conditions on Day 1 of each of 4 periods.
  Interventions: Drug: Mitapivat 100 mg; Drug: Placebo for Treatment B
- Treatment C (Experimental): Participants will receive a single oral dose of mitapivat 100 mg and placebo under high-fat meal conditions on Day 1 of each of 4 periods.
  Interventions: Drug: Mitapivat 100 mg; Drug: Placebo for Treatment C
- Treatment D (Experimental): Participants will receive a single oral dose of mitapivat 300 mg under fasted conditions on Day 1 of each of 4 periods.
  Interventions: Drug: Mitapivat 300 mg

INTERVENTIONS:
Drug: Placebo for Treatment A — 6 tablets matched to mitapivat tablet
  Arms: Treatment A
Drug: Mitapivat 100 mg — Two 50-mg tablets
  Other Names: AG-348
  Arms: Treatment B; Treatment C
Drug: Placebo for Treatment B — 4 tablets matched to mitapivat tablet
  Arms: Treatment B
Drug: Mitapivat 300 mg — Six 50-mg tablets
  Other Names: AG-348
  Arms: Treatment D
Drug: Placebo for Treatment C — 4 tablets matched to mitapivat tablet
  Arms: Treatment C

SUMMARY:
This is a Phase 1, randomized, single-dose, double-blinded, 4-period, crossover study to evaluate the pharmacokinetics, safety, and tolerability of mitapivat in healthy adult participants under fasted and fed (high-fat meal) conditions. Secondary objectives include evaluating the effect of mitapivat on electrocardiogram (ECG) parameters, including concentration-QT interval corrected for heart rate (C-QTc) analysis under fasted conditions. The study will include a 28-day screening period, four 7-day treatment periods. Participants will receive a follow-up telephone call within 28 (±1) days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participant is male or female 18 to 55 years of age, inclusive;
* If female, is not currently pregnant or breastfeeding OR is of non-childbearing potential, defined as either:

  * Being clinically infertile as the result of surgical sterilization, confirmed postmenopausal status, or another documented medical condition (eg, was born without a uterus) OR
  * Agreeing to either abstain from sexual intercourse with a male partner OR agrees to use a highly effective form of contraception, beginning at the time of screening and continuing throughout the study and for 28 days after dosing. The following are considered highly effective forms of contraception: hormonal oral contraceptives, injectables, and patches; intrauterine devices; double-barrier methods (synthetic condom, diaphragm, or cervical cap used with spermicidal foam, cream, or gel); and male partner sterilization;
* If male, agrees to abstain from sexual intercourse with a female partner OR agrees to use a highly effective form of contraception, beginning at the time of screening and continuing throughout the study and for 90 days after dosing, AND to refrain from donating sperm for the duration of the study and for 90 days after dosing;
* Participant has a body mass index 18 to 32 kilograms per square meter (kg/m^2), inclusive, at screening;
* Participant is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening;
* Participant has no clinically significant history or presence of ECG findings as judged by the investigator at screening and check-in, including each criterion as follows:

  * Normal sinus rhythm (heart rate [HR] between 45 beats per minute [bpm] and 100 bpm inclusive);
  * QT interval corrected for HR using Fridericia's formula (QTcF) ≤450 milliseconds (msec);
  * QRS interval ≤110 msec; and confirmed by manual over read if >110 msec;
  * PR interval between 120 and 220 msec;
* Participant agrees to comply with all protocol requirements;
* Participant is able to provide written informed consent.

Exclusion Criteria:

* Participant has any medical or surgical condition that, in the opinion of the investigator, could affect study drug absorption, distribution, metabolism, or excretion;
* Participant has undergone any major surgical procedure within the 3 months prior to screening;
* Participant has a history of any primary malignancy (including any melanoma or suspicious undiagnosed skin lesions), with the exception of in situ basal cell or squamous cell carcinomas of the skin, cervical carcinoma in situ, or other malignancies that have been curatively treated and for which the participant has displayed no evidence of disease within the 5 years prior to screening;
* Participant has glucose-6-phosphate-dehydrogenase deficiency;
* Participant has a known history or presence of liver disease.
* Participant has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), or human immunodeficiency virus (HIV) types 1 or 2 antibodies at screening;
* Participant has liver function tests including alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, and total bilirubin that are greater than the upper limit of normal at screening or check-in (results may be repeated once);
* Participant has platelet count or hemoglobin and hematocrit values that are below the lower limit of normal at screening or check-in (results may be repeated once);
* Participant has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at screening or before the first dose of study drug or throughout the study.
* Participant has used any prescription (excluding hormonal birth control) medications within 30 days (or 5 half-lives, whichever is longer) before the first dose of study drug or throughout the study;
* Participant has used any over-the-counter medications, including herbal or nutritional supplements, within 28 days (or 5 half-lives, whichever is longer) before the first dose of study drug or throughout the study;
* Participant has received study drug in another investigational study within 30 days (or 5 half-lives, whichever is longer) of dosing.
* Participant has donated blood or blood products >450 milliliters (mL) within 30 days before the first dose of study drug.
* Participant has history or presence of:

  * Risk factors for torsades de pointes (eg, heart failure, cardiomyopathy, or family history of long QT syndrome);
  * Sick sinus syndrome, second- or third-degree atrioventricular block, myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QT interval, or conduction abnormalities;
  * Repeated or frequent syncope or vasovagal episodes;
  * Hypertension, angina, bradycardia (if assessed as clinically significant by the investigator), or severe peripheral arterial circulatory disorders;
  * Clinically significant laboratory assessment findings, including hypokalemia, hypercalcemia, or hypomagnesemia;
* Participant has history or presence of:

  * Any evidence of atrial fibrillation, atrial flutter, complete right or left bundle branch block, or Wolff-Parkinson-White syndrome on the screening or baseline ECG;
  * Any morphology that renders measurement of QT interval imprecise (eg, neuromuscular artifact that cannot be readily eliminated, indistinct QRS onset, low-amplitude T-wave, merged T and U-waves, prominent U-waves, arrhythmia) on the screening or baseline ECG.
* Participant is not willing to refrain from marijuana or cannabinol-containing products for 7 days before the first dose of study drug and throughout the study;
* Participant has consumed caffeine- or xanthine containing products within 24 hours prior to first dose of study drug or throughout the study;
* Participant has consumed grapefruit or grapefruit juice, Seville orange or Seville orange containing products (eg, marmalade) within 28 days before the first dose of study drug or throughout the study;
* Participant has consumed fruit juices 72 hours prior to first dosing or during the study (with exception to the juices in relation to the fruits specified above);
* Participant has consumed vegetables from the mustard green family (eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussel sprouts, and mustard), or charbroiled meats for 7 days prior to first dose of study drug or throughout the study;
* Participant is a smoker or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, vaporizers, or inhalers) within 6 months before the first dose of study drug;
* Participant has a history of alcohol abuse or drug addiction within the last year or excessive alcohol consumption (regular alcohol intake >21 units per week for male participants and >14 units of alcohol per week for female participants) (1 unit is equal to approximately ½ pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits) or consumed alcohol 72 hours before the first dose of study drug or throughout the follow-up telephone call;
* Participant is involved in strenuous activity or contact sports within 24 hours before the first dose of study drug or throughout the study;
* Participant has a history of relevant drug and/or food allergies (ie, allergy to mitapivat or excipients [microcrystalline cellulose, croscarmellose sodium, sodium stearyl fumarate, magnesium stearate, and mannitol]);
* Participant has a history of allergy to sulfonamides (eg, co-trimoxazole antibiotic, silver sulfadiazine topical antibiotic for burn wounds) that has been characterized by acute hemolytic anemia, drug-induced liver injury, anaphylaxis, rash of erythema multiforme type, or Stevens-Johnson syndrome;
* In the opinion of the investigator, the participant is not suitable for entry into the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) From Time 0 to the Last Quantifiable Concentration (AUC0-T) for Mitapivat Under Fasted and High-Fat Meal Conditions | Predose and at various timepoints through 120 hours postdose within each 7-day period
AUC From Time 0 Extrapolated to Infinity (AUC0-Inf) for Mitapivat Under Fasted and High-Fat Meal Conditions | Predose and at various timepoints through 120 hours postdose within each 7-day period
Maximum Observed Plasma Concentration (Cmax) for Mitapivat Under Fasted and High-Fat Meal Conditions | Predose and at various timepoints through 120 hours postdose within each 7-day period
Time to Reach Maximum Observed Plasma Concentration (Tmax) for Mitapivat Under Fasted and High-Fat Meal Conditions | Predose and at various timepoints through 120 hours postdose within each 7-day period
Apparent Terminal Elimination Half-Life (T1/2) for Mitapivat Under Fasted and High-Fat Meal Conditions | Predose and at various timepoints through 120 hours postdose within each 7-day period
Apparent Oral Clearance (CL/F) for Mitapivat Under Fasted and High-Fat Meal Conditions | Predose and at various timepoints through 120 hours postdose within each 7-day period
Apparent Terminal Elimination Rate Constant (Λz) for Mitapivat Under Fasted and High-Fat Meal Conditions | Predose and at various timepoints through 120 hours postdose within each 7-day period
Apparent Volume of Distribution (Vd/F) for Mitapivat Under Fasted and High-Fat Meal Conditions | Predose and at various timepoints through 120 hours postdose within each 7-day period
Relative Bioavailability (Frel; AUC0-Inf [fed]/AUC0-Inf [fasted]) for Fed Treatment Following Administration of Mitapivat 100-mg Dose | Predose and at various timepoints through 120 hours postdose within each 7-day period

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to approximately 8 weeks
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the study drug.
Percentage of Participants with Abnormalities in Clinical Laboratory Findings | Up to approximately 8 weeks
  Clinical laboratory tests will include hematology, serum chemistry, and urinalysis.
Percentage of Participants With Abnormalities in Vital Sign Measurements | Up to approximately 8 weeks
  Vital sign measurements will include systolic and diastolic blood pressure, pulse rate, respiratory rate, and body temperature.
Percentage of Participants With Abnormalities in 12-lead Electrocardiogram (ECG) Results | Up to approximately 8 weeks
Percentage of Participants With Abnormalities in Physical Examination Findings | Up to approximately 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No